CLINICAL TRIAL: NCT02261753
Title: A Randomised Controlled Trial to Compare Seizure Remission Outcome Following Resective Surgery With or Without Prior Treatment With Ketogenic Diet in Children With Epilepsy the Result of Focal Cortical Dysplasia Type II
Brief Title: Evaluating Dietary Intervention Before surgicaL Treatment for Epilepsy
Acronym: EDIBLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study oversight committees unanimously decided to stop the study early on 26/07/2017 due to poor recruitment.
Sponsor: University College, London (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/0688
Record Dates: First submitted 2014-09-26; First posted 2014-10-10 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2014-10

CONDITIONS: Cortical Dysplasia
Keywords: epilepsy surgery, outcome, ketogenic diet, ortical dysplasia
MeSH Terms: conditions — Malformations of Cortical Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Classical ketogenic diet (Active Comparator): The KD is a high fat, low carbohydrate, low protein diet designed to mimic the effects of fasting on the body. It will be administered by calculation as per local standardised classical KD protocol with utilisation of long chain fat in a ratio of 2:1 to 4:1 carbohydrate and protein.
  Interventions: Dietary Supplement: Classical ketogenic diet
- B: No pretreatment (No Intervention): Following the decision to proceed to surgery, if randomised to this arm a date will be given for surgery as per routine clinical practice. No KD pre-treatment will be undertaken.

INTERVENTIONS:
Dietary Supplement: Classical ketogenic diet — A high fat low carbohydrate, low protein diet.
  Arms: A: Classical ketogenic diet

SUMMARY:
The investigators are undertaking the first European Randomised Controlled Trial (RCT) for epilepsy surgery in children with FCD type II, to prospectively evaluate the role of the KD prior to surgery in improving seizure outcome. The investigators will evaluate the role of KD as a disease-modifying treatment to achieve seizure control and improve neurodevelopment and quality of life. Children age 3 - 15 years with pharmacoresistant epilepsy believed to be the result of focal cortical dysplasia type II, considered to be surgically treatable, will be randomised to either receive 6m treatment presurgery with a ketogenic diet, or to proceed direct to surgery (no pretreatment). Primary outcome will be the time to achieve a period of 6 months of seizure freedom from the date of randomisation. Tissue resected at surgery will also be evaluated with regard to the degree of any methylation of DNA.

DETAILED DESCRIPTION:
Epilepsy surgery is now an accepted and effective management for individuals with drug resistant focal onset epilepsy in carefully selected candidates. This aside, only two RCTs have been performed in adults in temporal lobe epilepsy [1,2], and none in children . Malformations of cortical development are the most common pathology responsible for drug resistant focal epilepsy in childhood [3}. In retrospective studies, successful surgical resection resulting in seizure freedom in malformations of cortical development has been reported in 42-87% of cases [4], dependent on the series reviewed and the completeness of resection. Outcome is related to extent and completeness of resection, but the extent of tissue to be removed remains a challenge, especially in very young patients, where the limits of a lesion may be unclear and eloquent cortex may be involved.

FCD is one specific type of malformation, of localised areas of abnormal cortex that may be subdivided into I, II and III dependent on the pattern determined and cell types involved. This is by definition a histological diagnosis as was recently classified by the International League Against Epilepsy [5]. Specifically FCD type II can usually be suggested by characteristic changes on an MRI scan. These changes include increased cortical thickness, blurring of the cortical-white matter junction, increased signal on T2-weighted images, a radially oriented linear or conical transmantle strip of T2 hyperintensity, cortical thinning and localized brain atrophy. FCD type II may be subdivided histopathologically into IIa and IIb but it can be difficult to distinguish between the two radiologically.

The KD is a high fat diet with a proven efficacy in the treatment of drug resistant epilepsy in children [6]. An RCT performed in children aged 2-16 years diagnosed with drug resistant epilepsy utilising either a classical or medium chain triglyceride KD, demonstrated >50% reduction in seizures in 38% of participants after 3 months compared to 6% where there was no change in standard treatment, with no difference seen between the two diets [7,8]. A further RCT utilising a more relaxed approach of the KD, the modified Atkins diet, demonstrated similar results [9]. One open label study suggested particular efficacy in children with epilepsy due to FCD [10].

Clinical trials of epigenetic pharmacological treatment are promising and already have been approved for cancer [11]. Intriguingly, the most commonly used AED is valproic acid (VPA), in which histone deacetylase (HDAC) inhibitor activity was discovered in 2001 [12]. The HDAC antagonizing effect of VPA is, however, considerably low compared to second generation HDAC inhibitors suberoylanilide hydroxamic acid (SAHA, Zolinza, Vorinostat), LBH598 or Romidepsin [11]. Unfortunately, all HDAC inhibitors bear the risk of severe side effects when systemically administered during pregnancy. Nevertheless, there is also evidence that the epigenetic machinery can be modified by nutrition and dietary concepts [13]; such a dietary concept is the KD. Stimulus-induced DNA methylation changes have been identified in postnatal brain [14], thus it can be anticipated that DNA methylation modifications contribute to the molecular memory of postmitotic neurons also in the epileptogenic network. We propose that therapies such as the KD that are directly or indirectly targeting the epigenetic machinery could be helpful to prevent, delay or retard drug-resistant epilepsy.

Recent experimental data in an animal model has shown that the classical KD attenuates epigenetic chromatin modifications (i.e. DNA methylation), a master regulator for gene expression and functional adaptation of the cell, thereby modifying disease progression [15]. This hypothesis suggests that epigenetic mechanisms play a pivotal role in epileptogenesis and that seizures can by themselves induce epigenetic chromatin modifications, aggravating the epileptogenic condition [15].

We will conduct the first RCT for epilepsy surgery in children with FCD type II, to prospectively evaluate the role of the KD prior to surgery.

120 children aged 3 - 15 years with a diagnosis of Focal Cortical Dysplasia (FCD) type II a or b (with consistent MRI changes), treatment failure of at least two anti-epileptic drugs (AEDs) in controlling continuing seizures, with seizure semiology consistent with focal onset agreed to be surgically treatable through FCD resection and continuing seizures for less than 5 years, will be included in the trial after parental/ legal representative consent. Children will be excluded if they have a history of less than two seizures in 6 months prior to randomisation or they have previously used the Ketogenic diet (KD) or administration of the KD is medically contraindicated. Patients will be recruited from 19 participating European sites in 8 countries undertaking ketogenic diet and epilepsy surgery in children.

Participants will be followed-up for minimum 24 months/maximum 48 months (depending on the timing of randomisation) after randomisation. Primary outcome will be time to 6 month remission (i.e. the time to achieve a period of 6 months of seizure freedom from the date of randomisation). Tissue removed at surgery will be assessed for DNA methylation.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3 - 15 years;
2. MRI changes consistent with a diagnosis of FCD type II a or b;
3. History of at least two epileptic seizures in the past 6 months before randomisation;
4. Seizure semiology consistent with focal onset, agreed after pre-surgical discussion to be surgically treatable;
5. Parent/ legal representative willing to give consent.

Exclusion Criteria:

1. Previous use of the KD;
2. Not a surgical candidate for FCD resection;
3. Administration of the KD is medically contraindicated.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2014-10; Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Time to 6 month remission | Month 33
  the time to achieve a period of 6 months of seizure freedom from the date of randomisation pretreated KD group vs non pretreated group

SECONDARY OUTCOMES:
Time to first seizure from date of randomisation; | 33 months
  The time to first seizure from date of randomisation, KD pretreated vs non pretreated group
Time to 12 month remission after randomisation | 45 months
  Time to 12 month remission from seizures from date of randomisation, KD pretreated vs non pretreated group
Time to 24 month remission after randomisation (if enough time for follow-up is available) | 45 months
  Time to 24 months remission from seizures from date of randomisation, KD pretreated vs non pretreated group
Quality of life at 12 (and at 24 months if enough time for follow-up is available) | 45 months
  As determined by KINDL questionnaire, comparison of pretreated vs non pretreated group
Adaptive behaviour assessment at 12 months, after randomisation (and at 24 months if enough time for follow-up is available); | 45 months
  Comparison of neurodevelopmental change between pretreated and non pretreated KD group, as measured by Vineland adaptive behaviour scales
Methylation changes in tissue (DNA) from children pre-treated with the ketogenic diet compared to those not pretreated | 60 months
  As measured from tissue resected at surgery
Changes in peripheral DNA (blood platelets) following treatment with the KD | 60 months
  As measured from samples taken following the KD
Proportion of immediate AEs following resective surgery (i.e. surgical complications within 30 days) | 45 months
  As compared between groups, group pre-treated with KD compared to those without
Compare the general AE occurrence | 60 months
  As compared between groups, group pre-treated with KD compared to those without

CONTACTS AND LOCATIONS:
Overall Officials: J Helen Cross, MB ChB PhD, Principal Investigator — UCL-London
Locations (15):
- Johns Hopkins Hospital, Baltimore, Maryland, United States
- Medical University Vienna, Vienna, Austria
- Motol University Hospital, Prague, Czechia
- France (2):
  - Hospices Civil De Lyon, Lyon
  - Hopital de Hautepierre, Strasbourg
- Germany (2):
  - Krakenhaus Mara Maraweg, Bielefeld
  - Schpn Klinik Vogtareuth, Vogtareuth
- Italy (2):
  - Childrens Hospital Meyer, Florence
  - Ospedale Pediatric Bambino Gesu, Rome
- Hopitaux Universitaires de Geneve, Geneva, Switzerland
- United Kingdom (5):
  - Birmingham Childrens Hospital, Birmingham
  - Bristol Childrens Hospital, Bristol
  - Royal Hospital for Sick Children, Edinburgh
  - Great Ormond Street Hospital for Children NHS Trust, London
  - Manchester Childrens Hospital, Manchester

REFERENCES:
- [Background] Wiebe S, Blume WT, Girvin JP, Eliasziw M; Effectiveness and Efficiency of Surgery for Temporal Lobe Epilepsy Study Group. A randomized, controlled trial of surgery for temporal-lobe epilepsy. N Engl J Med. 2001 Aug 2;345(5):311-8. doi: 10.1056/NEJM200108023450501. PMID 11484687
- [Background] Engel J Jr, McDermott MP, Wiebe S, Langfitt JT, Stern JM, Dewar S, Sperling MR, Gardiner I, Erba G, Fried I, Jacobs M, Vinters HV, Mintzer S, Kieburtz K; Early Randomized Surgical Epilepsy Trial (ERSET) Study Group. Early surgical therapy for drug-resistant temporal lobe epilepsy: a randomized trial. JAMA. 2012 Mar 7;307(9):922-30. doi: 10.1001/jama.2012.220. PMID 22396514
- [Background] Harvey AS, Cross JH, Shinnar S, Mathern GW; ILAE Pediatric Epilepsy Surgery Survey Taskforce. Defining the spectrum of international practice in pediatric epilepsy surgery patients. Epilepsia. 2008 Jan;49(1):146-55. doi: 10.1111/j.1528-1167.2007.01421.x. Epub 2007 Nov 27. PMID 18042232
- [Background] Lerner JT, Salamon N, Hauptman JS, Velasco TR, Hemb M, Wu JY, Sankar R, Donald Shields W, Engel J Jr, Fried I, Cepeda C, Andre VM, Levine MS, Miyata H, Yong WH, Vinters HV, Mathern GW. Assessment and surgical outcomes for mild type I and severe type II cortical dysplasia: a critical review and the UCLA experience. Epilepsia. 2009 Jun;50(6):1310-35. doi: 10.1111/j.1528-1167.2008.01998.x. Epub 2009 Jan 21. PMID 19175385
- [Background] Blumcke I, Thom M, Aronica E, Armstrong DD, Vinters HV, Palmini A, Jacques TS, Avanzini G, Barkovich AJ, Battaglia G, Becker A, Cepeda C, Cendes F, Colombo N, Crino P, Cross JH, Delalande O, Dubeau F, Duncan J, Guerrini R, Kahane P, Mathern G, Najm I, Ozkara C, Raybaud C, Represa A, Roper SN, Salamon N, Schulze-Bonhage A, Tassi L, Vezzani A, Spreafico R. The clinicopathologic spectrum of focal cortical dysplasias: a consensus classification proposed by an ad hoc Task Force of the ILAE Diagnostic Methods Commission. Epilepsia. 2011 Jan;52(1):158-74. doi: 10.1111/j.1528-1167.2010.02777.x. Epub 2010 Nov 10. PMID 21219302
- [Background] Levy RG, Cooper PN, Giri P. Ketogenic diet and other dietary treatments for epilepsy. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001903. doi: 10.1002/14651858.CD001903.pub2. PMID 22419282
- [Background] Neal EG, Chaffe H, Schwartz RH, Lawson MS, Edwards N, Fitzsimmons G, Whitney A, Cross JH. The ketogenic diet for the treatment of childhood epilepsy: a randomised controlled trial. Lancet Neurol. 2008 Jun;7(6):500-6. doi: 10.1016/S1474-4422(08)70092-9. Epub 2008 May 2. PMID 18456557
- [Background] Neal EG, Chaffe H, Schwartz RH, Lawson MS, Edwards N, Fitzsimmons G, Whitney A, Cross JH. A randomized trial of classical and medium-chain triglyceride ketogenic diets in the treatment of childhood epilepsy. Epilepsia. 2009 May;50(5):1109-17. doi: 10.1111/j.1528-1167.2008.01870.x. Epub 2008 Nov 19. PMID 19054400
- [Background] Sharma S, Sankhyan N, Gulati S, Agarwala A. Use of the modified Atkins diet for treatment of refractory childhood epilepsy: a randomized controlled trial. Epilepsia. 2013 Mar;54(3):481-6. doi: 10.1111/epi.12069. Epub 2013 Jan 7. PMID 23294191
- [Background] Jung DE, Kang HC, Kim HD. Long-term outcome of the ketogenic diet for intractable childhood epilepsy with focal malformation of cortical development. Pediatrics. 2008 Aug;122(2):e330-3. doi: 10.1542/peds.2008-0012. PMID 18676519
- [Background] Hahnen E, Hauke J, Trankle C, Eyupoglu IY, Wirth B, Blumcke I. Histone deacetylase inhibitors: possible implications for neurodegenerative disorders. Expert Opin Investig Drugs. 2008 Feb;17(2):169-84. doi: 10.1517/13543784.17.2.169. PMID 18230051
- [Background] Gottlicher M, Minucci S, Zhu P, Kramer OH, Schimpf A, Giavara S, Sleeman JP, Lo Coco F, Nervi C, Pelicci PG, Heinzel T. Valproic acid defines a novel class of HDAC inhibitors inducing differentiation of transformed cells. EMBO J. 2001 Dec 17;20(24):6969-78. doi: 10.1093/emboj/20.24.6969. PMID 11742974
- [Background] Feil R, Fraga MF. Epigenetics and the environment: emerging patterns and implications. Nat Rev Genet. 2012 Jan 4;13(2):97-109. doi: 10.1038/nrg3142. PMID 22215131
- [Background] Feng J, Zhou Y, Campbell SL, Le T, Li E, Sweatt JD, Silva AJ, Fan G. Dnmt1 and Dnmt3a maintain DNA methylation and regulate synaptic function in adult forebrain neurons. Nat Neurosci. 2010 Apr;13(4):423-30. doi: 10.1038/nn.2514. Epub 2010 Mar 14. PMID 20228804
- [Background] Kobow K, Kaspi A, Harikrishnan KN, Kiese K, Ziemann M, Khurana I, Fritzsche I, Hauke J, Hahnen E, Coras R, Muhlebner A, El-Osta A, Blumcke I. Deep sequencing reveals increased DNA methylation in chronic rat epilepsy. Acta Neuropathol. 2013 Nov;126(5):741-56. doi: 10.1007/s00401-013-1168-8. Epub 2013 Sep 5. PMID 24005891